CLINICAL TRIAL: NCT02567318
Title: Is the Volume of the Caudate Nuclei Associated With Area of Secondary Hyperalgesia? - A Study of Healthy Volunteers
Brief Title: Is the Volume of the Caudate Nuclei Associated With Area of Secondary Hyperalgesia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Sejer Hansen, M.D., Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: SM3-MSH-2015
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Pain; Secondary Hyperalgesia; Healthy Volunteers; Magnetic Resonance Imaging
Keywords: Pain; Secondary hyperalgesia; Healthy volunteers; Magnetic Resonance Imaging
MeSH Terms: conditions — Pain; Hyperalgesia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI-scan (Experimental): All study participants will complete a MRI-scan of the brain
  Interventions: Device: MRI-scan

INTERVENTIONS:
Device: MRI-scan — Magnetic resonance imaging scan of the brain

SUMMARY:
The purpose of this prospective study is to investigate the degree of association between the volume of important pain-relevant structures in the brain and the size of the areas of secondary hyperalgesia.

DETAILED DESCRIPTION:
The healthy study participants will be included from the cohort of a previous study (NCT02527395) where areas of secondary hyperalgesia, heat pain detection thresholds, pain during 1 min. thermal stimulation and test results from the Pain Catastrophizing Scale and the Hospital Anxiety and Depression Score will be retrieved. The study consists of 1 study day. The study day will be conducted at a maximum of 2 months and a minimum of 2 weeks after the completion of the previous study (NCT02527395).The results of the previous study (NCT02527395) will be blinded until all participants have completed the study day.

All study participants will complete a MRI-scan of the brain.

The MRI scans will be performed with a Siemens MAGNETOM Verio 3 tesla, with b17 software, and a 32-channel head coil. The MRI-scan sequence is as follows:

* 3D Localiser
* 3D T1 weighted iso
* AX Diffusion tensor imaging
* AX Epi resting state fMRI
* AX Gre field map
* AX Epi ASL
* AX T2-weighted blade
* AX T2-weighted flair
* AX T2-weighted* Gre

Total MRI-scan time is estimated to approximately 40 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <35 years
* Speak and understand Danish
* Male sex
* Study participants who have understood and signed the informed consent
* No prescription medicine during the last 30 days.
* Have participated and completed the study with the identifier: NCT02527395.

Exclusion Criteria:

* Study participants that cannot cooperate to the test.
* Study participants who have a weekly intake of >21 units of alcohol, or a have consumed >3 units of alcohol within 24 hours before experimental day.
* Study participants with a substance abuse, assessed by the investigator.
* Study participants, who have consumed analgesics less than 3 days before experimental day.
* Study participants, who have consumed antihistamines less than 48 hours before experimental day.
* Study participants, who have consumed antidepressant medication during the last 30 days before experimental day.
* Study participants with chronic pain.
* Study participants with neurological illnesses.
* Study participants with psychiatric diagnoses.
* Study participants with a Body Mass Index of >30 kg/m2 or <18 kg/m2
* Study participants with Contraindications to MRI
* Study participants that decline information regarding potential pathological findings in relation to the MRI.
* Study participants that have any kind of trauma resulting in pain and administration of analgesics in the period between experimental pain testing and MRI-scan.
* Study participant that experience a head trauma in the period between the experimental pain testing and the MRI-scan.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Volume of the caudate nuclei, evaluated by mm3, and size of the area of secondary hyperalgesia following brief thermal sensitization, evaluated by cm2. | 40 minutes
  To investigate how close the volume of Caudate nucleus of the right and left hemisphere is associated with the size of the area of secondary hyperalgesia induced by Brief Thermal Sensitization.

SECONDARY OUTCOMES:
Volume of cortical and subcortical areas, evaluated by mm3, and size of the area of secondary hyperalgesia following brief thermal sensitization, evaluated by cm2. | 40 minutes
  To investigate the association between cortical and subcortical brain areas relevant for pain processing and the area of secondary hyperalgesia (Primary somatosensory cortex, anterior and mid Cingulate cortex, Basal ganglia (Putamen, Accumbens nucleus, and Globus pallidus), Insula, and the Cerebellum.
White matter microstructure, evaluated by tract based spatial statistics, and size of the area area of secondary hyperalgesia, evaluated by cm2 | 40 minutes
  By Diffusion Tensor Imaging to investigate the association between area of secondary hyperalgesia and white matter microstructure using tract based spatial statistics (TBSS).
White matter microstructure, evaluated by tract based spatial statistics, and size of the area area of secondary hyperalgesia, evaluated by cm2 | 40 minutes
  By Diffusion Tensor Imaging to conduct white-matter tractography to determine the connections between cortical and subcortical brain areas relevant for pain processing (Primary somatosensory cortex, anterior and mid Cingulate cortex, Basal ganglia (Putamen, Accumbens nucleus, and Globus pallidus), Insula, and the Cerebellum)

OTHER OUTCOMES:
Volume of the nucleus caudatus, evaluated by mm3, and heat pain detection threshold, registered by degrees celsius. | 40 minutes
  to investigate how close the volume of the Caudate nucleus of the right and left hemisphere is associated with the heat pain detection threshold.
Volume of the nucleus caudatus, evaluated by mm3, and pain during 1 min. thermal stimulation, evaluated by maximum on the visual analog scale, 0-100mm. | 40 minutes
  To investigate how close the volume of the Caudate nucleus of the right and left hemisphere is associated with the maximum visual analog score (0-100mm) during 1 min. thermal stimulation (45 degrees celsius) of the skin.
Volume of the nucleus caudatus, evaluated by mm3, and pain during 1 min. thermal stimulation, evaluated by area-under-the curve of the visual analog scale, 0-100mm. | 40 minutes
  To investigate how close the volume of the Caudate nucleus of the right and left hemisphere is associated with the area under the curve of the visual analog score (0-100mm) during 1 min. thermal stimulation (45 degrees celsius) of the skin.
Volume of the caudate nucleus, evaluated by mm3, and scores of the Pain Catastrophizing Scale. | 40 minutes
  To investigate how close the volume of Caudate nucleus of the right and left hemisphere is associated with the total score and subscores (rumination, magnification, and helplessness) of the Pain Catastrophizing Scale.
Volume of the caudate nucleus, evaluated by mm3, and scores of the Hospital Anxiety and Depression Scale. | 40 minutes
  To investigate how close the volume of Caudate nucleus of the right and left hemisphere is associated with the total score and subscores (Anxiety and Depression) of the Hospital Anxiety and Depression Scale.
Volume of regions of interest, evaluated by mm3, and size of the area of secondary hyperalgesia, evaluated by cm2. | 40 minutes
  To investigate structural differences (volume) following whole brain analyses as well as association with the size of the area of secondary hyperalgesia. When comparing healthy volunteers with a large vs. small area of secondary hyperalgesia following brief thermal sensitization defined by the upper and lower quartile.
Regions of interest, evaluated by tract based spatial statistics, and size of the area of secondary hyperalgesia, evaluated by cm2. | 40 min.
  To investigate differences in the association between area of secondary hyperalgesia and regions of interest extracted from tract based spatial statistics, when comparing healthy volunteers with a large vs. small area of secondary hyperalgesia following brief thermal sensitization defined by the upper and lower quartile.
Differences in white matter microstructure, evaluated by white-matter tractography. | 40 minutes
  To investigate differences in white matter microstructure in connections between pain related areas (Primary somatosensory cortex, anterior and mid Cingulate cortex, Basal ganglia (Putamen, Accumbens nucleus, and Globus pallidus), Insula, and the Cerebellum) evaluated by white-matter tractography, When comparing healthy volunteers with a large vs. small area of secondary hyperalgesia following brief thermal sensitization defined by the upper and lower quartile.
Differences in resting state network, evaluated by fMRI. | 40 minutes
  To investigate differences in resting state networks as investigated by resting state functional MRI by independent component analysis (dual regression method), when comparing healthy volunteers with a large vs. small area of secondary hyperalgesia following brief thermal sensitization defined by the upper and lower quartile.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansen MS, Asghar MS, Wetterslev J, Pipper CB, Johan Martensson J, Becerra L, Christensen A, Nybing JD, Havsteen I, Boesen M, Dahl JB. Is the Volume of the Caudate Nuclei Associated With Area of Secondary Hyperalgesia? - Protocol for a 3-Tesla MRI Study of Healthy Volunteers. JMIR Res Protoc. 2016 Jun 17;5(2):e117. doi: 10.2196/resprot.5680. PMID 27317630